CLINICAL TRIAL: NCT05197621
Title: The Impact of COVID-19 on Maternal and Neonatal Outcomes
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Integrated Research Center for Fetal Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00246472
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Pregnancy; Infection
MeSH Terms: conditions — COVID-19; Pregnancy Complications, Infectious | interventions — CVnCoV COVID-19 vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood, maternal breast milk, cord blood, neonatal blood, urine, and stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine Arm: Pregnant women who are planning to receive an mRNA COVID vaccine (Pfizer of Moderna), and/or a third booster vaccine, who consent to maternal blood collection before receipt of the vaccine and at 6 time points after receiving the vaccine and/or booster.
  Interventions: Biological: mRNA COVID-19 vaccine (Pfizer or Moderna)
- Sample Collection at Delivery Arm: Pregnant patients who have tested positive for COVID during their pregnancy or have a positive COVID test at the time of admission to Labor & Delivery, who consent to collection of maternal blood, cord blood, placenta, and breast milk samples, as well as neonatal blood and stool samples. Patients testing negative for COVID at the time of admission to Labor & Delivery can be enrolled in the study as controls.

INTERVENTIONS:
Biological: mRNA COVID-19 vaccine (Pfizer or Moderna) — mRNA vaccine received at any time during pregnancy course
  Other Names: Pfizer or Moderna COVID-19 vaccine
  Groups: Vaccine Arm

SUMMARY:
The novel coronavirus (SARS-CoV-2) infection (COVID-19) has caused a worldwide pandemic. There is still much that is unknown regarding the virus, especially its effects on pregnancy, the fetus, and the neonate. This study seeks to evaluate adverse pregnancy and neonatal outcomes related to COVID-19 infection.

The FDA has authorized emergency use authorization for the SARS-CoV-2 messenger ribonucleic acid (mRNA) vaccines from Pfizer and Moderna. Pregnant women were excluded from the Phase III clinical trials of the mRNA vaccines. There are no studies that have evaluated functional antibody responses, antibody reactivity to variant viruses, T cell frequencies or activity, or protection against infection or development of COVID-19. Having a more detailed understanding of how pregnancy and lactation alters the longevity, specificity, and activity of antiviral antibody and T cell-mediated immune responses to COVID-19 mRNA vaccines is essential for the FDA to inform future recommendations and regulation of these vaccines.

ELIGIBILITY:
Inclusion Criteria for Vaccine Arm:

* All pregnant women receiving their prenatal care from the Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center, who are planning to receive an mRNA COVID vaccine and/or a third dose booster during their pregnancy.

Exclusion Criteria:

* Prior COVID-19 infection.

Inclusion Criteria for Sample Collection Arm:

* All pregnant women admitted to the Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center for delivery and their newborn (at birth), will be considered for enrollment.
* Pregnant patients with a positive COVID-19 test during their pregnancy or at the time of admission to Labor & Delivery.

Exclusion Criteria:

* None

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female
Study Population: All pregnant women, aged 14-55, receiving prenatal care from Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center, who are planning to receive an mRNA COVID vaccine and/or a third dose booster during their pregnancy, or, patients who have had a positive COVID-19 test during their pregnancy or at the time of admission to Labor & Delivery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2028-05-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biospecimens from recently delivered pregnant women and neonates who were diagnosed with COVID-19 during their pregnancy | Testing will be performed from the time of study enrollment up to one year after sample collection
  Evaluation of biospecimens (maternal & neonatal blood, cord blood, placenta samples, neonatal stool samples & breast milk) collected from recently delivered pregnant women and neonates for biomarkers of placental inflammation and early onset neonatal sepsis.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of COVID-19 mRNA vaccines in pregnant and lactating people | Testing will be performed from the time of study enrollment up to one year after sample collection
  Investigation of antibody responses to COVID-19 mRNA vaccination in pregnant and lactating people over the course of one-year post vaccination (from both initial vaccine and booster administrations).
To evaluate the immunogenicity of COVID-19 mRNA vaccines in pregnant and lactating people | Testing will be performed from the time of study enrollment up to one year after sample collection
  Identification of T cell responses to COVID-19 mRNA vaccination in pregnant and lactating people over the course of one-year post vaccination (from both initial vaccine and booster administrations).
To evaluate the efficacy of COVID-19 mRNA vaccines in pregnant and lactating people | Testing will be performed from the time of study enrollment up to one year after sample collection
  Determination of SARS-CoV-2 vaccine efficacy and characterization of breakthrough infections with SARS-CoV-2 variants that evaded vaccine induced immunity.

CONTACTS AND LOCATIONS:
Overall Officials: William C Golden, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No